CLINICAL TRIAL: NCT05522998
Title: Efficacy and Safety of Ciprofol for the Induction of General Anesthesia in Obese Patients Undergoing Laparoscopic Sleeve Gastrectomy
Brief Title: Efficacy and Safety of Ciprofol in Laparoscopic Sleeve Gastrectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Third People's Hospital of Chengdu (Other)
Responsible Party: Principal Investigator, Xiaowei Chi, Principal Investigator, The Third People's Hospital of Chengdu
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022063
Record Dates: First submitted 2022-08-26; First posted 2022-08-31 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Bariatric Surgery
Keywords: Efficacy; Safety; Ciprofol; General anesthesia induction; Laparoscopic sleeve gastrectomy
MeSH Terms: interventions — (2-(1R)-1-cyclopropyl)ethyl-6-isopropyl-phenol; Propofol; Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ciprofol Group (Experimental): Experimental drug: Ciprofol; Dosage form: injection; Specification: 20ml: 50mg; Frequency and duration: intravenous infusion with micropump, anesthesia induction dose 0.4-0.5mg/kg, Administration for 30s (± 5S)
  Interventions: Drug: Ciprofol
- Propofol Group (Active Comparator): Experimental drug: Propofol; Dosage form: injection; Specification: 20ml: 200mg; Frequency and duration: intravenous infusion with micropump, anesthesia induction dose 2-2.5mg/kg, Administration for 30s (± 5S)
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Ciprofol — Ciprofol (0.4-0.5mg/kg) for anesthesia induction
  Other Names: Ciprofol Group; Experimental Group
  Arms: Ciprofol Group
Drug: Propofol — propofol(2-2.5mg/kg) for anesthesia induction
  Other Names: Propofol Group; Control Group
  Arms: Propofol Group

SUMMARY:
To evaluate the efficacy and safety of ciprofol for the induction of general anesthesia in obese patients undergoing laparoscopic sleeve gastrectomy. A randomized, parallel, propofol injection positive control study will be conducted to select obese patients who will undergo laparoscopic sleeve gastrectomy in the author's hospital. To evaluate the efficacy and safety, the main observation index, secondary observation indexes, safety evaluation indexes, and the incidence of postoperative adverse reactions will be recorded and compared between the two groups.

DETAILED DESCRIPTION:
To evaluate the efficacy and safety of ciprofol for the induction of general anesthesia in obese patients undergoing laparoscopic sleeve gastrectomy. A randomized, parallel, propofol injection positive control study will be conducted to select obese patients who will undergo laparoscopic sleeve gastrectomy in the author's hospital. To evaluate the efficacy and safety, the following indexes will be recorded and compared between the two groups.

* The main observation index：(1) The rate of successful anesthesia induction
* Secondary observation indexex：(1) Time from initial administration of study drug to loss of consciousness; (2) Time from initial administration of study drug to disappearance of eyelash reflex; (3) Changes in bispectral index(BIS) values during anesthesia induction
* Safety evaluation indexes：(1) Adverse events; (2) Intubation response rate; (3) Vital signs; (4) Evaluation of injection pain
* Adverse events to be focused on：(1)The incidence of blood pressure reduction requiring treatment during anesthesia induction; (2) The incidence of respiratory depression

ELIGIBILITY:
Inclusion Criteria:

* 18 < age ≤ 65, regardless of gender;
* ASA is classified as grade I-III;
* BMI≥35kg/m2
* Obese patients who need laparoscopic sleeve gastrectomy under general anesthesia;
* The subjects voluntarily participated in the trial and signed the informed consent.

Exclusion Criteria:

* Contraindications to general anesthesia;
* Accompanied by infectious heart disease such as myocarditis or endocarditis, septicemia;
* Brain injury, possible intracranial hypertension, cerebral aneurysm, cerebrovascular accident history and central nervous system diseases: mental system diseases (schizophrenia, mania, insanity, etc.) and long-term history of taking psychotropic drugs, or other diseases that hinder the measurement of BIS value;
* Acute heart failure, unstable angina pectoris, myocardial infarction within 6 months before screening, resting ECG heart rate ≤ 50 beats / min, third degree atrioventricular block and other serious arrhythmias, serious heart valve disease, QTc: male ≥ 450ms, female ≥ 470ms;
* Abnormal liver and kidney function (ALT or AST ≥ 2.5 times the upper limit of normal value, TBIL ≥ 1.5 times the upper limit of normal value), abnormal renal function (bun or urea ≥ 1.5 times the upper limit of normal value, cr> the upper limit of normal value, or dialysis treatment within 28 days before operation), or obvious abnormal coagulation function (pt/ aptt/tt higher than the upper limit of normal value), anemia or thrombocytopenia (HB ≤ 90g/l, PLT ≤ 80 × 109/L)
* Those whose blood pressure was not satisfactorily controlled (SBP ≥ 160mmhg and / or DBP ≥ 100 mmHg in sitting position during screening period);
* SBP in sitting position during screening period ≤ 90mmHg;
* Diabetes subjects whose blood glucose was not satisfactorily controlled (fasting blood glucose ≥ 11.1mmol/l in the screening period and / or random blood glucose ≥ 13.6 mmol/l);
* Have a history of drug abuse and alcoholism within 2 years before the screening period. Alcoholism is defined as regular drinking for more than 14 times / week (once =150 ml wine or 360 ml beer or 45 ml spirits);
* The subjects who were judged to have difficulty in respiratory management were rated as grade IV by modified Mahalanobis score;
* Known or suspected allergy or contraindication to various components of the study drug or other benzodiazepines, opioids, propofol, muscle relaxants, etc;
* Pregnant or lactating women or subjects with birth plan within 6 months (including men);
* Those who participated in any clinical trial as subjects within 3 months before enrollment;
* Other circumstances determined by the researcher as unsuitable for inclusion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
The rate of successful anesthesia induction | Through study completion, an average of 1 year
  The criteria for success are to meet the following two requirements at the same time: 1) successful induction (i.e. improved investigator awake / sedation score (MOAA / S) ≤ 1) after the administration of the study drug (at most 2 additional times are allowed); 2) No alternative anesthetics were used.

SECONDARY OUTCOMES:
Time to LOC | During anesthesia induction, an average of 10 minutes
  Time from initial administration of study drug to loss of consciousness
Time to disappearance of eyelash reflex | During anesthesia induction, an average of 10 minutes
  Time from initial administration of study drug to disappearance of eyelash reflex
BIS | During anesthesia induction, an average of 10 minutes
  Changes in bispectral index(BIS) values during anesthesia induction

CONTACTS AND LOCATIONS:
Overall Officials: Xiaowei Chi, M.D., Principal Investigator — Third People's Hospital of Chengdu, Southwest Jiaotong University
Locations (1):
- The Third People's Hospital of Chengdu, Affiliated Hospital of Southwest Jiaotong University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chi X, Xu Y, Li Q, Xia K, Fu Q. Efficacy and safety of ciprofol for the induction of general anesthesia in patients with obesity undergoing laparoscopic sleeve gastrectomy: A double-blind randomized, controlled study. PLoS One. 2025 Jul 24;20(7):e0329005. doi: 10.1371/journal.pone.0329005. eCollection 2025. PMID 40705792